CLINICAL TRIAL: NCT05720598
Title: Staging LaParoscopy to Assess Lymph NOde InvoLvement in Advanced GAstric Cancer - POLA Study
Brief Title: Staging LaParoscopy to Assess Lymph NOde InvoLvement in Advanced GAstric Cancer
Acronym: POLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Collaborators: Ohio State University (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POLA
Record Dates: First submitted 2023-01-19; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Gastric Cancer; Lymph Node Metastasis
Keywords: Gastric Cancer; ICG; Staging Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis | interventions — Gastroscopy; Indocyanine Green; Injections

STUDY DESIGN:
Intervention Model Description: Patients with histopathologically confirmed, locally advanced adenocarcinoma of the stomach scheduled for staging laparoscopy by the multidisciplinary team will be classified for enrollment into this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients underdoing staging laparoscopy with indocyanine green (ICG) (Experimental): Patients will undergo upper GI endoscopy one day before SL will be dissolved in sterile water, resulting in a 0.125mg/ml concentration. 2 milliliters of the solution will be injected into the submucosa of 4 peritumoral sites - 0.5ml for each site. The following day patient will undergo SL
  Intraoperative application of ICG-enhanced vision will be accomplished with dedicated optical devices. Alternate usage of white light and ICG fluorescence mode will allow precise location and cT stage determination of primary tumor, followed by identification of SN and its corresponding LN station, according to Japanese Gastric Cancer Association guidelines. Identified SN will be retrieved with a high-energy device, and the LN basin will be labeled with a magnetic clip.
  Interventions: Procedure: Sentinel Node Assessment; Procedure: Staging laparoscopy; Procedure: Gastroscopy with indocyanine green (ICG) injection

INTERVENTIONS:
Procedure: Sentinel Node Assessment — The SN assessment will be conducted similarly to the method proposed by Märkl et al. All LNs will be stored in a -80 °C freezer, immediately after retrieval. Within 1 to 3 days, each LN will be individually measured and weighed. Small LNs (<5 mm in short diameter) will be bisected, and half of the node will be processed for histological evaluation while the remaining half will be used for OSNA analysis. For intermediate-sized LNs (5-10 mm), a middle slice of about 2 mm thickness will be cut out for the histology, and the remaining parts of the node will be processed by OSNA. In large LNs (>10 mm), at least two slices will be cut out for histology, and the remaining parts of the node will be analyzed by OSNA.
Procedure: Staging laparoscopy — Pneumoperitoneum (10-12mmHg) will be obtained with Veress needle or 10mm trocar after minilaparotomy. Peritoneal cavity will be thoroughly assessed after insertion of two additional trocars. In cases of macroscopic dissemination, peritoneal cancer index (PCI) will be determined. After switching the optical camera into near-infrared / indocyanine green fluorescence mode, the primary tumor will be visualized, followed by assessment and possible dissection of sentinel lymph node with a high-energy device. The lymph node will be retrieved with a sterile bag, and the area of dissection will be marked with a clip. Trocars will be removed under visual assistance, and the pneumoperitoneum will be released through trocars in order to prevent port-site metastases.
Procedure: Gastroscopy with indocyanine green (ICG) injection — Patients will undergo gastroscopy one day prior to staging laparoscopy. The ICG powder contains 0.125 mg/ml. Two milliliters of ICG (0.125mg/ml) solution is injected in the submucosa with into four peritumoral sites, 0.5 ml for each site.

SUMMARY:
Staging LaParscopy to Assess Lymph NOde InvoLvement in Advanced GAstric Cancer (POLA) study aims to investigate the safety and feasibility of ICG-guided SN retrieval in GC patients undergoing multimodal treatment. The pretreatment clinical variables potentially associated with the procedure will also be analyzed.

To the best of our knowledge, the current study is the first to evaluate the role of ICG in SN biopsy in advanced GC patients undergoing multimodal treatment.

DETAILED DESCRIPTION:
Comprehensive lymph node assessment seems to be critical for proper treatment strategy and survival prediction, particularly in advanced GC. Recent data on the sentinel node (SN) concept in early GC has shown favorable results regarding LN detection rate and clinical status determination. Staging laparoscopy (SL) with lavage cytology provides an additional value to the clinical staging of GC, particularly in detecting occult peritoneal disease. The role of Indocyanine green (ICG) guided SN mapping in GC confirmed its technical feasibility. ICG can be safely used to identify SN, determine the surgical resection line, improve the LN harvest, and reduce noncompliance in patients undergoing D2 lymphadenectomy.

The majority of the studies focused on the aspect of the increase in LN harvest. At the same time, no data exist regarding its potential role in GC nodal staging. To the best of our knowledge, the current study is the first to evaluate the role of ICG in SN biopsy in advanced GC patients undergoing multimodal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed gastric adenocarcinoma (or undifferentiated carcinoma)
3. Stage II - III disease (cT2-4a, N0-3, M0) based on the pretreatment CT and 8th edition of TNM classification
4. Qualification for SL by the decision of the multidisciplinary tumor board
5. Written informed consent for endoscopy and SL

Exclusion Criteria:

1. Early GC (cT1N0-3M0) scheduled for endoscopic treatment by the multidisciplinary tumor board
2. Previous abdominal surgery which could interfere lymphatic basin of the stomach, including previous gastrectomy, endoscopic (sub)mucosal dissection
3. Distant metastasis (cM1) clinically apparent in pretreatment abdominal/pelvic CT
4. Technical inability to perform endoscopic ICG injection or ICG injection beyond the submucosa
5. Visual inability to identify the SN during SL
6. Positive cytology (cyt+) after SL
7. Other malignancies
8. History of allergy to iodine agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the identification rate of ICG-guided SN in advanced GC patients. | Up to 2 weeks after inclusion in the study, during staging laparoscopy
  The identification rate will allow confirmation of the safety and feasibility of ICG-guided SN biopsy during staging laparosocpy in advanced GC patients

SECONDARY OUTCOMES:
Pathological status of the retrieved sentinel node | Up to 2 weeks after staging laparoscopy
  SN retrieved during staging laparoscopy will undergo microscopic evaluation. The histopathological report will contain information on the character of the lymph node (benign/metastatic)
Pathological status and regression grade of the retrieved sentinel node after neoadjuvant chemotherapy | Up to 2 weeks after gastrectomy, 1 month after completion of neoadjuvant chemotherapy and 3 months after initial staging laparoscopy
  SN retrieved during gastrectomy will undergo microscopic evaluation. The histopathological report will contain information on the character of the lymph node (benign/metastatic) and its regression grade according to Becker classification

CONTACTS AND LOCATIONS:
Overall Officials: Karol Rawicz-Pruszyński, MD,PhD, Principal Investigator — Department of Surgical Oncology, Medical University of Lublin, Poland
Locations (1):
- Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rawicz-Pruszynski K, Sedlak K, Pelc Z, Mlak R, Litwinski J, Manko P, Zinkiewicz K, Pasnik I, Cieszczyk K, Pawlik T, Markl B, Erodotou M, Polkowski WP. Staging LaParoscopy to Assess Lymph NOde InvoLvement in Advanced GAstric Cancer (POLA)-Study protocol for a single-arm prospective observational multicenter study. PLoS One. 2023 May 19;18(5):e0285758. doi: 10.1371/journal.pone.0285758. eCollection 2023. PMID 37205666